CLINICAL TRIAL: NCT06585982
Title: Gut Microbiota Profile Analysis and Randomized Controlled Trials (RCT) Study of the Effect of Synbiotics on Insulin and TNF-α in Metabolic Dysfunction -Associated Fatty Liver Disease (MAFLD)
Brief Title: Synbiotics Impact on Insulin and TNF-α in MAFLD: a Gut Microbiota Profile Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Diponegoro (Other)
Collaborators: Dr. Kariadi General Hospital Medical Center (Other); PT Kalbe Farma Tbk (Industry)
Responsible Party: Principal Investigator, Adriyan Pramono, Lecturer, Universitas Diponegoro
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-1583
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Fatty Liver Disease
Keywords: Metabolic dysfunction-associated fatty liver disease; Gut Microbiota; Metabolic profile; Synbiotic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Drug coding and group assignment are done by the pharmacy, where the investigator only receives data in the form of sample coding but does not know whether the coded sample received an intervention or control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RILLUS (Active Comparator): Treatment group receive RILLUS, a synbiotic that each tablet contains Viable cells 1.0 x 109 CFU containing three types of prebiotic species (Lactobacillus plantarum 8.55mg, Streptococcus thermophilus 8.55mg, and Bifidobacterium bifidum 2.55 mg) and Fructooligosaccharide (FOS) 480 mg as prebiotic.
  Interventions: Dietary Supplement: Treatment
- Placebo (Placebo Comparator): Control group receive what appeared to be RILLUS, but only placebo containing Fructooligosaccharide, Xylitol DC, Isomalt, Microcrystalline cellulose, Corn starch, Milk flavor powder, Hydroxypropyl methylcellulose, Vanilla flavor powder, Magnesium stearate
  Interventions: Dietary Supplement: Control

INTERVENTIONS:
Dietary Supplement: Treatment — RILLUS is a synbiotic produced by Kalbe Farma
  Arms: RILLUS
Dietary Supplement: Control — Placebo produced by Kalbe Farma
  Arms: Placebo

SUMMARY:
Primary Objective: To analyze the effect of synbiotic supplementation on metabolic profile, insulin and TNF-α and gut microbiota changes in patients with Metabolic dysfunction-Associated Fatty Liver Disease (MAFLD).

Research question: Are there any changes in metabolic profile, Insulin and TNF-α and gut microbiota changes in MAFLD patients after synbiotic supplementation

Participants will:

* Treatment group given supplementation and the control group will be given placebo at a dose of 2x1 tablet for 12 weeks.
* Patients will visit the hospital every 28 days for up to 4 months for control and follow-up supplementation.
* patients will be given a supplement consumption compliance logbook and a food record logbook used to record food consumption filled in by the patient.

DETAILED DESCRIPTION:
Non-alcoholic Fatty Liver Disease (NAFLD) is a common chronic liver disease estimated to affect 25% of the global population. NAFLD is defined as the presence of fat in the liver that is not associated with alcohol consumption. The researchers proposed a new term, Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD), which covers a range of liver conditions associated with metabolic dysregulation, including obesity and type 2 diabetes. MAFLD is a systemic disease with complications such as obesity, which is closely related to glucose and lipid metabolism. Obesity is associated with comorbidities such as dyslipidaemia, hypertension and diabetes.

The pathogenesis mechanism of MAFLD is complex and involves several factors such as mitochondrial dysfunction, oxidative stress, and increased free fatty acids (FFA). The 'multi-hit' theory explains how lifestyle, environmental and genetic factors contribute to the development of MAFLD. The gut microbiota also plays an important role in the development of MAFLD through the gut-liver axis, where microbiota imbalance can lead to inflammation and liver damage.

Research shows the microbiota composition in MAFLD patients is different from healthy people, with an increase in Proteobacteria and Actinobacteria and a decrease in butyrate-producing bacteria. Interventions with probiotics and prebiotics (synbiotics) have been shown to reduce liver fibrosis and improve metabolic profiles. The investigators are interested in assessing the effects of synbiotics on changes in metabolic biomarkers, insulin, TNF-α, and gut microbiota in MAFLD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged 25-55 years
2. Patients are willing to become research respondents after filling out informed consent
3. Patients can and are willing to consume supplements orally within a predetermined time
4. Patients are willing to record compliance with taking supplements in a diary that has been provided
5. Patients diagnosed with MAFLD by FibroScan interpreted by a specialist in gastroenterology-hepatology with a CAP score ≥263 dB/m

Exclusion Criteria:

1. Patients with hepatitis (hepatitis B, hepatitis C, and autoimmune hepatitis) and alcoholic liver disease, cirrhosis of the liver
2. Patients who are pregnant, or breastfeeding or in a programme to become pregnant during participation in this study.
3. Patients with a history of alcohol consumption >40 g/day.
4. Patients with a history of decompensated disease including ascites, encephalopathy, variceal haemorrhage
5. Patients with Hepatocellular Carcinoma (HCC)
6. Patients with a history of bowel resection or bariatric surgery Patients with chronic inflammatory bowel disease (IBD)
7. Patients with a history of antibiotic use or probiotic/prebiotic/synbiotic consumption in the past 1 month
8. Use of Vitamin E and omega-3 fatty acids
9. Patients who were not hospitalised in the last month and therefore did not have any food restrictions related to their illness.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2025-03-07 (Estimated); Study Completion 2025-03-07 (Estimated)

PRIMARY OUTCOMES:
Complete Hematology | 3 months
  Complete Hematology analysis before and after intervention
Metabolic Profile | 3 months
  Analyzing fasting glucose and HbA1C before and after the intervention
Metabolic Profile | 3 months
  Analyzing liver function SGOT (Serum Glutamic Oxaloacetic Transaminase) and SGPT (Serum Glutamic Pyruvic Transaminase) before and after intervention
Metabolic Profile | 3 months
  Analyzing lipid profile (total cholesterol, triglycerides, HDL, LDL) before and after intervention
Insulin | 3 months
  Insulin test results were taken before and after the intervention
TNF-alpha | 3 months
  TNF-alpha test results were taken before and after the intervention
CRP (C-Reactive Protein) | 3 months
  Analyzing C-Reactive Protein (CRP) before and after intervention

SECONDARY OUTCOMES:
Alpha Diversity of Gut Microbioata | 4 months
  Calculation of Gut Microbiota's species diversity index using Shannon Index, where the gene expresion were observed at OTUs level.
Anti-HCV | 3 months
  Anti-HCV test is used as a screening to ensure respondents do not have hepatitis
HBsAg (Hepatitis B Surface Antigen) | 3 months
  HBsAg test is used as a screening to ensure respondents do not have hepatitis
Beta Diversity of Gut Microbioata | 4 months
  Calculation of Gut Microbiota's species diversity index using Bray Curtis, where the gene expresion were observed at OTUs level.

CONTACTS AND LOCATIONS:
Overall Officials: Hery D Purnomo, Dr, Principal Investigator — Dr. Kariadi Medical Hospital
Locations (1):
- RSUP Dr. Kariadi, Semarang, Semarang, Indonesia

IPD SHARING:
Plan to Share IPD: No
Based on the consent from the respondent that already written in inform consent, we cannot legally give the information to anyone else

REFERENCES:
- [Background] Meagratia, R. A., Cayami, F. K., Bahrudin, U., Lestari, W., Maharani, N., Faradz, S. M., & Purnomo, H. D. (2021). Adiponutrin and Adiponectin Gene Variants in Indonesian Patients with Non-Alcoholic Fatty Liver Disease: a Preliminary Study. In Journal of Biomedicine and Translational Research (Vol. 7, Issue 2, pp. 86-91). Institute of Research and Community Services Diponegoro University (LPPM UNDIP). https://doi.org/10.14710/jbtr.v7i2.11777
- [Background] Verma N, Duseja A, Mehta M, De A, Lin H, Wong VW, Wong GL, Rajaram RB, Chan WK, Mahadeva S, Zheng MH, Liu WY, Treeprasertsuk S, Prasoppokakorn T, Kakizaki S, Seki Y, Kasama K, Charatcharoenwitthaya P, Sathirawich P, Kulkarni A, Purnomo HD, Kamani L, Lee YY, Wong MS, Tan EXX, Young DY. Machine learning improves the prediction of significant fibrosis in Asian patients with metabolic dysfunction-associated steatotic liver disease - The Gut and Obesity in Asia (GO-ASIA) Study. Aliment Pharmacol Ther. 2024 Mar;59(6):774-788. doi: 10.1111/apt.17891. Epub 2024 Feb 1. PMID 38303507
- [Background] The Relationship between the Duration of Suffering from Diabetes and HbA1c Levels with the Degree of Liver Stiffness in Type 2 Diabetes Mellitus Patients
- [Background] Byrne CD, Targher G. NAFLD: a multisystem disease. J Hepatol. 2015 Apr;62(1 Suppl):S47-64. doi: 10.1016/j.jhep.2014.12.012. PMID 25920090
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Background] Boccatonda A, Andreetto L, D'Ardes D, Cocco G, Rossi I, Vicari S, Schiavone C, Cipollone F, Guagnano MT. From NAFLD to MAFLD: Definition, Pathophysiological Basis and Cardiovascular Implications. Biomedicines. 2023 Mar 13;11(3):883. doi: 10.3390/biomedicines11030883. PMID 36979861
- [Background] Eslam M, Newsome PN, Sarin SK, Anstee QM, Targher G, Romero-Gomez M, Zelber-Sagi S, Wai-Sun Wong V, Dufour JF, Schattenberg JM, Kawaguchi T, Arrese M, Valenti L, Shiha G, Tiribelli C, Yki-Jarvinen H, Fan JG, Gronbaek H, Yilmaz Y, Cortez-Pinto H, Oliveira CP, Bedossa P, Adams LA, Zheng MH, Fouad Y, Chan WK, Mendez-Sanchez N, Ahn SH, Castera L, Bugianesi E, Ratziu V, George J. A new definition for metabolic dysfunction-associated fatty liver disease: An international expert consensus statement. J Hepatol. 2020 Jul;73(1):202-209. doi: 10.1016/j.jhep.2020.03.039. Epub 2020 Apr 8. PMID 32278004
- [Background] Mathews SE, Kumar RB, Shukla AP. Nonalcoholic steatohepatitis, obesity, and cardiac dysfunction. Curr Opin Endocrinol Diabetes Obes. 2018 Oct;25(5):315-320. doi: 10.1097/MED.0000000000000432. PMID 30074500
- [Background] Rachmatullah TF, Permatadewi CO, Hutami HT, Limantoro C, Purnomo, MD, PhD HD. Correlation between Non-Alcoholic Fatty Liver Disease (NAFLD) fibrosis score (NFS) with Left Ventricular Mass Index (LVMI) in patients with NAFLD. J Biomed Transl Res. 2021 Aug 31;7(2):79-85.
- [Background] Purnomo HD, Kasno, Sudijanto E, Hirlan, Darmono, Daldiyono, et al. The roles of metabolic syndrome and several biomarkers in incidence and severity of non-alcoholic fatty liver disease. Hiroshima J Med Sci. 2018;67(4):138-46.
- [Background] Buzzetti E, Pinzani M, Tsochatzis EA. The multiple-hit pathogenesis of non-alcoholic fatty liver disease (NAFLD). Metabolism. 2016 Aug;65(8):1038-48. doi: 10.1016/j.metabol.2015.12.012. Epub 2016 Jan 4. PMID 26823198
- [Background] Tilg H, Adolph TE, Moschen AR. Multiple Parallel Hits Hypothesis in Nonalcoholic Fatty Liver Disease: Revisited After a Decade. Hepatology. 2021 Feb;73(2):833-842. doi: 10.1002/hep.31518. Epub 2021 Feb 6. No abstract available. PMID 32780879
- [Background] Boursier J, Diehl AM. Nonalcoholic Fatty Liver Disease and the Gut Microbiome. Clin Liver Dis. 2016 May;20(2):263-75. doi: 10.1016/j.cld.2015.10.012. Epub 2015 Dec 24. PMID 27063268
- [Background] Park E, Jeong JJ, Won SM, Sharma SP, Gebru YA, Ganesan R, Gupta H, Suk KT, Kim DJ. Gut Microbiota-Related Cellular and Molecular Mechanisms in the Progression of Nonalcoholic Fatty Liver Disease. Cells. 2021 Oct 2;10(10):2634. doi: 10.3390/cells10102634. PMID 34685614
- [Background] Zhang Y, Yan S, Sheng S, Qin Q, Chen J, Li W, Li T, Gao X, Wang L, Ang L, Ding S. Comparison of gut microbiota in male MAFLD patients with varying liver stiffness. Front Cell Infect Microbiol. 2022 Aug 3;12:873048. doi: 10.3389/fcimb.2022.873048. eCollection 2022. PMID 35992168
- [Background] Oh JH, Lee JH, Cho MS, Kim H, Chun J, Lee JH, Yoon Y, Kang W. Characterization of Gut Microbiome in Korean Patients with Metabolic Associated Fatty Liver Disease. Nutrients. 2021 Mar 21;13(3):1013. doi: 10.3390/nu13031013. PMID 33801023
- [Background] Behrouz V, Aryaeian N, Zahedi MJ, Jazayeri S. Effects of probiotic and prebiotic supplementation on metabolic parameters, liver aminotransferases, and systemic inflammation in nonalcoholic fatty liver disease: A randomized clinical trial. J Food Sci. 2020 Oct;85(10):3611-3617. doi: 10.1111/1750-3841.15367. Epub 2020 Sep 4. PMID 32885440
- [Background] Bomhof MR, Parnell JA, Ramay HR, Crotty P, Rioux KP, Probert CS, Jayakumar S, Raman M, Reimer RA. Histological improvement of non-alcoholic steatohepatitis with a prebiotic: a pilot clinical trial. Eur J Nutr. 2019 Jun;58(4):1735-1745. doi: 10.1007/s00394-018-1721-2. Epub 2018 May 19. PMID 29779170
- [Background] Mofidi F, Poustchi H, Yari Z, Nourinayyer B, Merat S, Sharafkhah M, Malekzadeh R, Hekmatdoost A. Synbiotic supplementation in lean patients with non-alcoholic fatty liver disease: a pilot, randomised, double-blind, placebo-controlled, clinical trial. Br J Nutr. 2017 Mar;117(5):662-668. doi: 10.1017/S0007114517000204. Epub 2017 Mar 27. PMID 28345499